CLINICAL TRIAL: NCT00629018
Title: The Effects of Autologous Intracoronary Stem Cell Transplantation In Patients With End-Stage Dilated Cardiomyopathy
Brief Title: Safety and Efficacy Study of Stem Cell Transplantation to Treat Dilated Cardiomyopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Blood Transfusion Centre of Slovenia (Other Government); Stanford University (Other)
Responsible Party: Principal Investigator, Bojan Vrtovec, prof. dr. Bojan vrtovec, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DCM-SCT1
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Dilated Cardiomyopathy
Keywords: Stem Cells; Heart Failure; Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SC Group (Experimental): SC therapy,'Bone Marrow Stimulation','CD34+ autologous stem cell transplantation':
  In the SC group, CD34+ cells were mobilized by granulocyte colony-stimulating factor and collected via apheresis. Patients underwent myocardial scintigraphy and cells were injected in the artery supplying segments with the greatest perfusion defect
  Interventions: Biological: CD34+ autologous stem cell transplantation; Drug: Bone Marrow Stimulation; Biological: SC therapy
- Controls (No Intervention): Patients receiving no cell therapy.

INTERVENTIONS:
Biological: CD34+ autologous stem cell transplantation — Peripheral blood stem cells will be mobilized by daily subcutaneous injections of filgrastim; CD34+ cells will be collected via apheresis and labeled with technetium. Patients will undergo myocardial perfusion scintigraphy for myocardial viability assessment and the collected CD34+ cells will be injected intracoronary in the artery supplying the segments of reduced tracer accumulation
  Arms: SC Group
Drug: Bone Marrow Stimulation — Patients will undergo filgrastim stimulation and viability assessment using the same protocol as in Arm 1. However, in this group, no intracoronary stem cell delivery will be performed; the patients will receive placebo (saline).
  Other Names: G-CSF stimulation
  Arms: SC Group
Biological: SC therapy — In the SC group, CD34+ cells were mobilized by granulocyte colony-stimulating factor and collected via apheresis. Patients underwent myocardial scintigraphy and cells were injected in the artery supplying segments with the greatest perfusion defect
  Arms: SC Group

SUMMARY:
Several studies have documented that transplantation of bone marrow-derived cells (BMC) following acute myocardial infarction is associated with a reduction in infarct scar size and improvements in left ventricular function and perfusion. The available evidence in humans suggests that BMC transplantation is associated with improvements in physiologic and anatomic parameters in both acute myocardial infarction and chronic ischemic heart disease, above and beyond the conventional therapy. In particular, intracoronary application of BMC is proved to be safe and was associated with significant improvement in the left ventricular ejection fraction (LVEF) in patients with chronic heart failure.

In contrast to ischemic heart failure, the data on effects of BMC transplantation in patients with dilated cardiomyopathy are limited to pre-clinical studies. In a rat model of dilated cardiomyopathy, intramyocardial delivery of pluripotent mesenchymal cells improved LVEF, possibly through induction of myogenesis and angiogenesis, as well as by inhibition of myocardial fibrosis, suggesting that the beneficial effects of stem cell transplantation in dilated cardiomyopathy may primarily be related to their ability to supply large amounts of angiogenic, antiapoptotic, and mitogenic factors. Similarly, transplantation of cocultured mesenchymal stem cells and skeletal myoblasts was shown to improve LVEF in a murine model of Chagas disease.

Study Aim:

To define the clinical effects of BMC transplantation in dilated cardiomyopathy in a pilot clinical study investigating the effects of intracoronary CD34+ cell transplantation on functional, structural, neurohormonal, and electrophysiologic parameters in patients with end-stage dilated cardiomyopathy.

DETAILED DESCRIPTION:
Patients were randomly allocated in a 1:1 ratio to receive intracoronary transplantation of autologous CD34+ stem cells (SC group) or no intracoronary infusion (control group). At the time of enrollment, and at yearly intervals thereafter, we performed detailed clinical evaluation, echocardiography, 6-minute walk test, and measured plasma levels of NT-proBNP. To better-define the potential role of inflammatory response, we also measured plasma inflammatory markers (tumor necrosis factor [TNF]-α and interleukin [IL]-6) at the time of CD34+ stem cell injection.

ELIGIBILITY:
Inclusion Criteria:

* Normal coronary angiogram
* Left ventricular ejection fraction < 40%
* NYHA III or IV heart failure symptoms
* Bone marrow reactivity (G-CSF test)
* Presence of viable myocardium

Exclusion Criteria:

* Hematologic malignancy
* Multiorgan failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2006-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Torre Amione, MD, PhD, Study Director — Methodist DeBakey Heart Center, Houston TX, USA; Francois Haddad, MD, Study Director — Stanford University
Locations (1):
- Ljubljana University Medical Center, Ljubljana, Slovenia

REFERENCES:
- [Derived] Vrtovec B, Poglajen G, Sever M, Lezaic L, Domanovic D, Cernelc P, Haddad F, Torre-Amione G. Effects of intracoronary stem cell transplantation in patients with dilated cardiomyopathy. J Card Fail. 2011 Apr;17(4):272-81. doi: 10.1016/j.cardfail.2010.11.007. Epub 2010 Dec 24. PMID 21440864

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of an open-label randomized study design conducted at the Advanced Heart Failure and Transplantation Center at University Medical Center Ljubljana in collaboration with the Methodist DeBakey Heart Center and Stanford University.
Pre-assignment Details: Patients with acute multi-organ failure or history of haematologic neoplasms were not included.
Groups:
- SC Group: 55 patients were randomized to CD34+ cell transplantation (SC group). In the SC group, peripheral CD34+cells were mobilized by G-CSF and collected via apheresis. Patients underwent myocardial scintigraphy and CD34+ cells were injected in the artery supplying the segments with reduced viability
- Control Group: 55 patients were randomized to standard medical therapy, without stem cell injection.
Period: Overall Study
Arm/Group | SC Group | Control Group
Started | 55 | 55
Completed | 55 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SC Group | Control Group | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 52 | 105
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (8) | 55 (7) | 54 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 45 | 44 | 89
Region of Enrollment [Number; unit: participants]
  Slovenia | 55 | 55 | 110

OUTCOME MEASURES:

1. Primary Outcome: Heart Failure Mortality
Time Frame: 5 years
Population: The minimal sample size for the study was calculated using a pre-specified power of 90% and P value of 0.05.
Measure: Number; unit: participants
Arm/Group | SC Group | Control Group
Number analyzed (Participants) | 55 | 55
participants | 8 | 19
Statistical Analysis 1: Comparison: SC Group vs Control Group; The minimal sample size for the study was calculated using a pre-specified power of 90% and P value of 0.05; Test type: Superiority or Other; p = 0.01, Log Rank

2. Primary Outcome: Changes in Left Ventricular Ejection Fraction
Description: Left ventricular ejection fraction measured by echocardiography
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: Percentage of ejection
Arm/Group | SC Group | Control Group
Number analyzed (Participants) | 55 | 55
Percentage of ejection
  Baseline | 24.3 (6.5) | 25.7 (4.1)
  5 years | 30.0 (5.1) | 23.3 (4.2)

3. Secondary Outcome: Changes in Exercise Capacity
Time Frame: 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Changes in Electrophysiologic Properties of Ventricular Myocardium
Time Frame: 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Changes in Plasma Inflammatory Markers
Time Frame: 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Changes in Left Ventricular Function
Time Frame: 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | SC Group | Control Group
Serious Adverse Events (participants affected / at risk) | 8/55 | 19/55
Other Adverse Events (participants affected / at risk) | 2/55 | 0/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SC Group (N=55) | Control Group (N=55)
Death (Cardiac disorders) | 8 | 19
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SC Group (N=55) | Control Group (N=55)
Non-sustained ventricular tachycardia (Cardiac disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes